CLINICAL TRIAL: NCT00671047
Title: The Systemic Lupus Erythematosus (SLE) Activity Gene Expression (SAGE) Study
Acronym: SAGE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: XDx (Industry)
Responsible Party: Debbie Pieretti, XDx, Inc.
Other Study IDs: SL105
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-12

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Autoimmune Diseases; Lupus
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: SLE subjects with flares in the last 12 months in specific organ systems.
  Interventions: Other: non-interventional

INTERVENTIONS:
Other: non-interventional — SLE nature history observational

SUMMARY:
The goal of this study is to enable the study sponsor to develop a new blood test method for clinicians to accurately predict which individuals with lupus will flare, when the flare will occur, and flare severity. Ultimately such a newly derived test would allow treating physicians to start pre-emptive therapy early, with the goal of achieving remission quickly and with a shorter duration of treatment; identify individuals who will have less severe flares and will thus require less aggressive treatments; or intensify and lengthen treatment for those individuals who will need such therapy.

The design of this study is to follow individuals with a known diagnosis of SLE for changes in disease activity during the course of one year of observation. Clinical data and blood and urine samples will be collected at scheduled monthly visits. The clinical data and blood samples will be used for identifying gene expression profile(s) that are associated with increases in SLE disease activity (lupus "flares").

DETAILED DESCRIPTION:
This study is currently enrolling individuals who have an established diagnosis of SLE to participate. There is no cost to volunteers who participate and the study pays for the visits to the clinics for monthly collection of clinical information and blood and urine samples. Women who are or become pregnant may participate in the study with the recommendation of their health care providers and the study doctors.

ELIGIBILITY:
Inclusion Criteria:

* Individual has met the diagnostic criteria for SLE (at least 4 out of the 11) American College of Rheumatology (ACR) criteria and:
* Has experienced specific manifestations of lupus disease activity within the last 12 months including the following:

  * Lupus nephritis (kidney disease); vasculitis and or central nervous system involvement and/or:
  * Required treatment with at least 20 mg per day of prednisone (or equivalent) and/or:
  * Required hospitalization directly due to SLE disease

Exclusion Criteria:

* Subjects unable or unlikely to cooperate with the procedures of the protocol
* Substance abuse / dependence that in the opinion of the investigator could compromise the subject's ability to complete the study
* Subject with a more dominant autoimmune disease, e.g. Rheumatoid arthritis, Sjogren's syndrome, multiple sclerosis, scleroderma
* History of malignancy within the last five years with the exception of basal cell carcinoma
* Active infection: Known HIV positive status, currently active tuberculosis , active infection receiving antibiotics
* Had tissue or organ transplantation (including bone marrow)
* On chronic hemo- or peritoneal dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2007-12; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: James Yee, MD, Ph.D., Study Director — XDx, Inc.
Locations (12):
- United States (11):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - East Bay Rheumatology Medical Group, San Leandro, California
  - Emory University, Atlanta, Georgia
  - Kansas University Medical Center, Kansas City, Kansas
  - State University of New York, Brooklyn, New York
  - North Shore Long Island Jewish Health System, Lake Success, New York
  - New York University, New York, New York
  - Hospital for Special Surgery, New York, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Metroplex Clinical Research Center, Dallas, Texas
- Toronto Western Hospital, Toronto, Ontario, Canada